CLINICAL TRIAL: NCT02989402
Title: A Prospective, 16 Week, Phase IV Study to Evaluate Safety, Tolerability and Effectiveness in Patients With Severe Dementia of the Alzheimer's Type Exposed to Rivastigmine (Exelon)15cm2 Transdermal Patch
Brief Title: A Phase IV Study to Evaluate Safety, Tolerability and Effectiveness of Rivastigmine Patch 15cm2 in Patients With Severe Dementia of the Alzheimer's Type.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CENA713DIN01
Record Dates: First submitted 2016-12-08; First posted 2016-12-12 (Estimated); Results first posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2023-12

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer, Rivastigmine
MeSH Terms: conditions — Alzheimer Disease | interventions — Rivastigmine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rivastigmine patch (Experimental): 15 cm^2 patch sizes loaded with 27 mg of rivastigmine - one patch per day
  Interventions: Drug: Rivastigmine

INTERVENTIONS:
Drug: Rivastigmine — 15 cm^2 patch sizes loaded with 27 mg of rivastigmine - one patch per day

SUMMARY:
This was a multicenter, prospective, phase IV study evaluating safety, tolerability and effectiveness of rivastigmine 27 mg -15 cm^2 transdermal patch prescribed in patients with severe dementia of the Alzheimer's type as per discretion of treating physician.

DETAILED DESCRIPTION:
This was a multicenter, prospective, single-arm, open-label, phase IV study to evaluate safety, tolerability and effectiveness of Rivastigmine 27 mg -15 cm^2 transdermal patch prescribed in patients with severe dementia of the Alzheimer's type as per discretion of treating physician. Male and female patients who were treated according to local routine clinical practice were enrolled in the study upon signing informed consent. The prescription decision was independent of the decision for inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing to participate in the study by providing written informed consent.
2. Patients diagnosed with severe dementia secondary to Alzheimer's disease (AD) 3 .Patient's prescribed with rivastigmine 27mg -15 cm^2 transdermal patch as per discretion of treating physician

Exclusion Criteria:

1. Contraindication as per PI
2. Patients simultaneously participating in other studies
3. Use of other investigational drugs within 5 half-lives of enrollment, or within 30 days (for small molecules) /until the expected PD effect has returned to baseline (for biologics)], whichever is longer.
4. History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- India (7):
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Banglaore, Karnataka
  - Novartis Investigative Site, Bengaluru, Karnataka
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
  - Novartis Investigative Site, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 9 investigative sites in India.
Pre-assignment Details: Participants who were treated according to local routine clinical practice were enrolled in the study upon signing informed consent.
Period: Overall Study
Arm/Group | Rivastigmine Patch
Started | 100
Completed | 72
Not Completed | 28
Not completed — Adverse event, or serious adverse event | 4
Not completed — Death | 2
Not completed — Discontinuation of study treatment and premature patient withdrawal | 3
Not completed — Lost to Follow-up | 8
Not completed — Patient no longer on monotherapy | 1
Not completed — Patient stopped Exelon® patch treatment | 1
Not completed — Withdrawal by Subject | 7
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | Rivastigmine Patch
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.3 (9.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 49
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with treatment emergent AEs (any AE regardless of seriousness), AEs related to study treatment, AEs led to study treatment discontinuation, and SAEs.
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment, plus 30 days post treatment, up to a maximum duration of approximately 142 days.
Population: The safety set included all patients who provided informed consent to collect information and who were treated with at least one patch of Rivastigmine 27 mg -15 cm2 transdermal patch during this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivastigmine Patch
Number analyzed (Participants) | 100
Participants
  At least one AE | 32
  AEs related to study treatment | 13
  AEs leading to treatment discontinuation | 4
  At least one SAE | 4

2. Secondary Outcome: Change From Baseline in Mini-Mental State Examination (MMSE)
Description: The MMSE is a brief, practical screening test for cognitive dysfunction. The test consists of five sections (orientation, registration, attention-calculation, recall, and language); and results in a total score can range from 0 to 30, with higher scores indicating better function.
Time Frame: Baseline, 16 weeks
Population: Patients in the intend to treat (ITT) set who had a valid assessment of the outcome measure at week 16. The intend to treat (ITT) set included all patients who signed the informed consent and who had at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Rivastigmine Patch
Number analyzed (Participants) | 63
Score on a scale | 3.1 (4.79)

3. Secondary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study - Activities of Daily Living Inventory - Severe Impairment Version (ADCS-ADL SIV) Score
Description: Alzheimer's Disease Cooperative Study - Activities of Daily Living Inventory - Severe Impairment Version (ADCS-ADL SIV) score is a tool to assess the ability of patients with moderate to severe dementia to perform activities of daily living. The ADCS-ADL SIV assessment is done at start and end of visit. The assessment includes 19 questions. The total score ranges from 0 - 54. Higher scores indicate less functional impairment and greater competence.
Time Frame: Baseline, 16 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Rivastigmine Patch
Number analyzed (Participants) | 69
Score on a scale | -1.6 (10.47)

4. Secondary Outcome: Compliance by Caregiver Medication Questionnaire (CMQ) Score
Description: Caregiver evaluation of the medications used for Alzheimer Disease was assessed using the Caregiver Medication Questionnaire (CMQ). Compliance was rated on a scale from 0 = "never took the medication as prescribed" to 10 = "always took the medication as prescribed."
Time Frame: Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Rivastigmine Patch
Number analyzed (Participants) | 69
Score on a scale | 8.1 (2.78)

5. Secondary Outcome: Number of Participants With a Skin Irritation
Description: The following score system were used to assess skin irritation:
  I. Dermal response:
  Score 0 = No erythema (normal skin) Score 1 = Erythema barely visible Score 2 = Mild erythema Score 3 = Moderate erythema Score 4 = Severe erythema Score 5 = Severe erythema with vesicles or blisters
Time Frame: Week 16
Population: Patients in the safety set who had a dermal response score at week 16. The safety set included all patients who provided informed consent to collect information and who were treated with at least one patch of Rivastigmine 27 mg -15 cm2 transdermal patch during this study.
Measure: Number; unit: participants
Arm/Group | Rivastigmine Patch
Number analyzed (Participants) | 70
participants
  Score 0 | 65
  Score 1 | 3
  Score 2 | 2
  Score 3 to 5 | 0

6. Secondary Outcome: Number of Participants With a Urinary Tract Infection (UTI)
Description: Urine samples were collected to assess the number of patients with UTI.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rivastigmine Patch
Number analyzed (Participants) | 100
Participants | 10

7. Secondary Outcome: Patch Adhesion to the Skin
Description: Patch adhesion to the skin was evaluated by the caregiver. An estimate of the patch adherence was provided and graded according to the patch adhesiveness score.
  Following scores were used to capture comments relating to patch adhesion:
  0 = 90 % adhered (essentially no lift off of the skin)
  1. = 75% to < 90% adhered (some edges only lifting off of the skin)
  2. = 50% to < 75% adhered (less than half of the patch lifting off the skin)
  3. = < 50% adhered but not detached (more than half the system lifting off of the skin without falling off)
  4. = the patch was completely detached. The score ranges from 1 to 4 where a higher score indicates less adhesion.
Time Frame: Week 16
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Rivastigmine Patch
Number analyzed (Participants) | 70
participants
  Score 0 | 60
  Score 1 | 4
  Score 2 | 0
  Score 3 | 4
  Score 4 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment, plus 30 days post treatment, up to a maximum duration of approximately 142 days.
Arm/Group | Rivastigmine Patch
All-Cause Mortality (participants affected / at risk) | 2/100
Serious Adverse Events (participants affected / at risk) | 4/100
Other Adverse Events (participants affected / at risk) | 16/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivastigmine Patch (N=100)
ARRHYTHMIA (Cardiac disorders) | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1
CEREBROSPINAL FLUID LEAKAGE (Nervous system disorders) | 1
DEMENTIA (Nervous system disorders) | 1
HYPONATRAEMIC SEIZURE (Nervous system disorders) | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivastigmine Patch (N=100)
VOMITING (Gastrointestinal disorders) | 3
URINARY TRACT INFECTION (Infections and infestations) | 10
DECREASED APPETITE (Metabolism and nutrition disorders) | 3
SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/02/NCT02989402/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT02989402/SAP_001.pdf